CLINICAL TRIAL: NCT00901940
Title: Single Centre Open-Label Randomised Trial of Meningococcal Serogroup ACYW-135 B Cell Response to Primary & Booster Doses of ACWY Conjugate Vaccine & Primary Dose of ACWY Polysaccharide With Booster Dose of ACWY Conjugate in Adults
Brief Title: Understanding the Immune Response to Meningitis Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Professor Andrew Pollard, Chief Investigator, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007/04
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-06

CONDITIONS: Meningitis; Septicemia
MeSH Terms: conditions — Meningitis; Sepsis | interventions — MenACWY; Meningococcal Vaccines; meningococcal group A polysaccharide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MenACWY Plain Polysaccharide (ACWY Vax) (Active Comparator): The MenACWY Plain Polysaccharide Vaccine, which is already licensed and is used as a travel vaccine, is known as the MenACWY plain polysaccharide (ACWY Vax). Participants in this arm will receive 1 dose of the MenACWY plain polysaccharide (ACWY Vax) and 1 dose of the MenACWY conjugate (MenACWY).
  Interventions: Biological: Meningococcal polysaccharide A, C, Y and W135 and Menveo
- MenACWY conjugate (Active Comparator): The MenACWY conjugate vaccine was licensed in the UK in March 2010, and is known as the MenACWY conjugate vaccine (Menveo). Participants in this arm will receive 2 doses of the MenACWY conjugate vaccine.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Conjugate

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Conjugate — 2 x 0.5 mL dose
  Other Names: MenACWY; Menveo
  Arms: MenACWY conjugate
Biological: Meningococcal polysaccharide A, C, Y and W135 and Menveo — 1 x 0.5 mL dose of ACWY Vax, 1 x 0.5 mL dose of Menveo
  Other Names: ACWY Vax; Menveo
  Arms: MenACWY Plain Polysaccharide (ACWY Vax)

SUMMARY:
The purpose of the study is to evaluate and compare the immune response to two vaccines against 4 related bacteria: meningococcal serogroups A, C, W-135 and Y. These bacteria can cause meningitis and /or septicaemia (blood poisoning). The two vaccines are a protein-polysaccharide conjugate vaccine (MenACWY)and a meningococcal plain polysaccharide vaccine(MenACWY PS). Both vaccines are licensed and are currently used for travellers to areas with a high incidence of invasive meningococcal disease. However, plain polysaccharide vaccines are known to be poorly immunogenic in children and they do not stimulate immunological memory, apart from the serogroup A component. In contrast, a protein-polysaccharide conjugate vaccine against meningococcal serogroups A, C, W-135 and Y has been found to be immunogenic in infants and to be able to induce immunological memory.

The proposed study is a single centre, open-label, randomised, controlled study in 150 healthy adults aged 18-70 years. The participants will be given either 2 injections of the meningococcal protein-polysaccharide conjugate vaccine one month apart, or one injection of the meningococcal plain polysaccharide vaccine followed one month later with an injection of the meningococcal conjugate vaccine. Blood samples will be collected before immunisation and at several time points following immunisations to evaluate the level of meningococcal specific antibody induced by two different vaccination regimes. The data derived from the study will be relevant in determining which of these vaccines should be used in preference in travellers who are receiving immunisation against meningococcal disease before travelling to high risk areas. Additionally, a number of scientific questions regarding the nature of the immune response to the two vaccines (specifically looking at the white blood cells responsible for producing antibodies, known as B cells) and the role of genetic variations in influencing the vaccine recipient's immune response will be addressed in the study.

DETAILED DESCRIPTION:
In this single centre, open-label, randomised, controlled study of 150 healthy adults aged 18-70 years we will be evaluating the immune response to immunisation with 2 different vaccines against 4 related bacteria known as Neisseria meningitidis serogroups A, C, W-135 and Y. These bacteria (also known as meningococci) can produce meningitis and septicaemia (blood poisoning). The first vaccine, which has been used as a travel vaccine in the UK for several years, is known as the MenACWY plain polysaccharide (MenACWY PS). The other vaccine, known as the MenACWY conjugate vaccine (MenACWY) was licensed in the UK in March 2010 and is now recommended as a travel vaccine by the Department of Health.

In order to evaluate the immune response to these vaccines we will be measuring not only the blood levels of antibodies specific to serogroup A, C, W-135 and Y meningococci, but also the population of white blood cells known as B cells which produce these antibodies. Two forms of these B cells will be measured, the plasma cells (which actively produce antibodies) and memory B cells (which do not produce antibodies but persist in the body and can be stimulated to turn into plasma cells when required).

Participants will be randomised into group I or group II on a 1:1 basis to receive either MenACWY or MenACWY PS. One month later, all participants will receive a booster dose of the MenACWY conjugate vaccine. The ACWY polysaccharide vaccine will be administered subcutaneously, and the MenACWY conjugate vaccine will be given intramuscularly. Each participant will be observed for at least 15 minutes after vaccination for any immediate reactions.

Blood samples will be collected from each participant for analysis prior to each immunisation, 7 days following the first immunisation and 7 and 28 days following the second immunisation. The volume of blood samples obtained at each timepoint will be 20 mLs. Blood will be used for antibody analysis (by ELISA), B cell analysis (by ELISpot)and DNA extraction for genetic analysis.

In summary, participants enrolled in this study will have a total of 5 visits in a period of 2 months. They will receive two doses of the MenACWY conjugate vaccine or one dose of the ACWY polysaccharide vaccine followed by one dose of the MenACWY conjugate vaccine. During this period they will have a total of 5 blood samples taken (5x20mL= 100 mL of blood taken in a 2 month period).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation after the nature of the study has been explained
* Male or Female, aged 18- 70 years inclusive
* In good health as determined by:

  * Medical history
  * History-directed physical examination
  * Clinical judgment of the investigator
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

* Are unwilling or unable to give written informed consent to participate in the study
* Have previously received any meningococcal vaccine (this will be confirmed with the participant's general practitioner after enrolment)
* Have previously been diagnosed with laboratory confirmed meningococcal disease
* Have a history of any anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component
* Have a known or suspected autoimmune disease or impairment /alteration of immune function resulting from (for example):

  * Receipt of any immunosuppressive therapy
  * Congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months or long-term systemic corticosteroid therapy* (*prednisolone or equivalent for more than two consecutive weeks within the past 3 months).
* Have a suspected or known HIV infection or HIV related disease
* Have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months
* Have a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time
* Have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* Participation in another clinical trial investigating a vaccine, a drug, a medical device, or a medical procedure
* Pregnancy as confirmed by a positive pregnancy test
* Currently breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be whether the SBA GMT at day 7 following MenACWY is ≥ 30% greater than that observed at day 7 following MenACWY PS. | Day 7

SECONDARY OUTCOMES:
The measurement of meningococcal serogroup C SBAs (using human complement) at day 7 following the initial immunisation with MenACWY and MenACWY PS. | Day 7
The measurement of meningococcal serogroup A and C specific SBAs (using human complement) at day 28 following the initial immunisation with MenACWY and MenACWY PS, and at day 7 and day 28 following the 'follow up' immunisation with MenACWY. | Day 7-28
Meningococcal serogroup W-135 and Y SBAs will also be performed on a subset of samples obtained at the above timepoints. | Day 7-28
The measurement of meningococcal serogroup A, C, W-135 and Y specific memory B cells and plasma B cells at day 7, and memory B cells at day 28 after first immunisation with MenACWY and MenACWY PS, and after the 'follow up' immunisation with MenACWY. | Day 7-56
Other assessments of the immune response to MenACWY and MenACWY PS (e.g. measurement of meningococcal serogroup A, C, W-135 and Y specific IgG by ELISA) may also be performed. | Day 7-56

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, FRCPCH, PhD, Principal Investigator — University of Oxford, Department of Paediatrics
Locations (1):
- University of Oxford, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, United Kingdom

REFERENCES:
- [Background] Ramasamy MN, Clutterbuck EA, Haworth K, Bowman J, Omar O, Thompson AJ, Blanchard-Rohner G, Yu LM, Snape MD, Pollard AJ. Randomized clinical trial to evaluate the immunogenicity of quadrivalent meningococcal conjugate and polysaccharide vaccines in adults in the United kingdom. Clin Vaccine Immunol. 2014 Aug;21(8):1164-8. doi: 10.1128/CVI.00099-14. Epub 2014 Jun 25. PMID 24964805